CLINICAL TRIAL: NCT05014724
Title: CIDP07 Rozanolixizumab Post Trial Access Program (the PTA)
Status: No longer available | Type: Expanded Access
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: CIDP07
Record Dates: First submitted 2021-08-19; First posted 2021-08-20 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Keywords: Chronic inflammatory demyelinating polyradiculoneuropathy; CIDP; UCB7665; rozanolixizumab
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — rozanolixizumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Rozanolixizumab — Rozanolixizumab is dosed weekly. Patients should continue to receive the dose they were receiving in the CIDP04 (NCT04051944) trial.

SUMMARY:
This Post Trial Access (PTA) Program enables access to rozanolixizumab for eligible patients who have taken part in the CIDP04 trial (NCT04051944) and are continuing to derive benefit from treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has taken part in the CIDP04 (NCT04051944) study
* Patient who derives continued benefit from treatment
* All required safety information has been reported as per local laws/regulations, reported to Bionical, as appropriate, and documented in the patient's medical records
* Patient is not pregnant

Exclusion Criteria:

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)